CLINICAL TRIAL: NCT05580380
Title: Addressing Health Disparities in Chronic Low Back Pain With Patient-Clinician Relatedness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-00141
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Chronic Low-Back Pain
Keywords: Patient-Clinician Relationship; Back Pain; Chronic Pain; Biopsychosocial; Health Disparities
MeSH Terms: conditions — Back Pain; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Limited Patient-Clinician Relationship Group (Active Comparator)
  Interventions: Other: Limited Relationship
- Enhanced Patient-Clinician Relationship Group (Experimental)
  Interventions: Other: Enhanced Relationship

INTERVENTIONS:
Other: Limited Relationship — In this group, participants will share information regarding their low back pain history to a clinician who is not providing eye-contact, has farther physical distance, and is not directly facing the participant. The clinician will not provide verbal affirmations or ask clarifying questions about the patient's low back pain history. Instead, more time will be spent on completion of documentation.
  Arms: Limited Patient-Clinician Relationship Group
Other: Enhanced Relationship — A condition in which the clinician is providing enhanced relatedness with consistent eye contact, closer physical distance, facing the patient, and providing non-verbal affirmations (i.e. nodding, smiling), as the participant shares their low back pain history. The clinician will provide empathic verbal affirmations and will ask clarifying questions about the patient's low back pain history.
  Arms: Enhanced Patient-Clinician Relationship Group

SUMMARY:
The primary objective of the current research is to assess the effect of an enhanced patient-clinician relationship when compared to a limited patient-clinician relationship on measures of chronic low back pain and objective functional measures.

The second objective is to examine racialized disparities in chronic low back pain among individuals who identify as non-Hispanic Black and non-Hispanic White using a qualitative approach.

Lastly, the study team will explore relationships between psychosocial components of low back pain, pain and functional outcomes, and patient-clinician relationship measures.

ELIGIBILITY:
Inclusion Criteria:

1. Self-reported low back pain located between the 12th rib and the gluteal fold.
2. Low back pain lasting at least 3-months.
3. Low back pain for more than half of the days in the past 6-months.
4. Age 18-45 years old.
5. Reports at least 3 out of 10 average pain over the past week on the numerical pain rating scale.
6. Reports having more back pain when compared to leg pain.

Exclusion Criteria:

1. Does not meet any of the above inclusion criteria.
2. If there is a reported low back procedure scheduled within the upcoming 8-weeks including an epidural injection or spinal surgery.
3. If low back pain care (i.e. physicians visits, physical therapy) is being received through Worker's Compensation or No Fault insurance.
4. Dizziness, vestibular, or visual difficulties that cause balance problems over the past 2-weeks.
5. Any lower or upper extremity surgery within the past year or any prior history of spine surgery, spinal fracture, or malignancy in the spine will not be included in the study.
6. Individuals who are pregnant or breastfeeding.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Number of lifts completed in 1 minute | Pre-Intervention (Day 1), Post-Intervention (Day 1)
  To be measured during the 1-minute lift test, where the participant is asked to lift objects of a certain weight.
Change in time holding the horizontal position | Pre-Intervention (Day 1), Post-Intervention (Day 1)
  To be collected during the Biering-Sorensen Test, which is a timed measure used to assess the endurance of the trunk extensor muscles.
Change in Trunk Flexion Range of Motion | Pre-Intervention (Day 1), Post-Intervention (Day 1)
  To be measured during the Fingertip-to-floor (FTF) Test, where the participant is asked to bed forward and attempt to reach the floor with their fingertips.
Change in Mean Walking Speed | Pre-Intervention (Day 1), Post-Intervention (Day 1)
  To be measured/assessed during the 4-meter walking test.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) for Pain | Pre-Intervention (Day 1), Post-Intervention (Day 1)
  VAS will be used to report pain at rest. A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 100 mm horizontal line, and this rating is then measured from the left edge (=VAS score). The total score range is 0 (no pain) to 10 (worst pain imaginable); the higher the score, the worse the pain.
Pain pressure threshold | Pre-Intervention (Day 1), Post-Intervention (Day 1)
  Pain pressure threshold (the degree of pressure required to produce symptoms) will be assessed using a pressure algometer.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Stolfi, PT, DPT, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Department of Physical Therapy, Arthur J. Nelson Human Performance Laboratory, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasongle request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to Angela.Stolfi@nyulangone.org. To gain access, data requestors will need to sign a data access agreement

REFERENCES:
- [Derived] Vorensky M, Squires A, Jones S, Sajnani N, Castillo E, Rao S. Impact of Patient-Clinician Relationships on Pain and Objective Functional Measures for Individuals with Chronic Low Back Pain: An Experimental Study. J Health Care Poor Underserved. 2024;35(4):1229-1257. doi: 10.1353/hpu.2024.a943987. PMID 39584210